CLINICAL TRIAL: NCT03376477
Title: A Randomized, Double-blind, Placebo-Controlled Phase II Trial of an Allogeneic Myeloma GM-CSF Vaccine With Lenalidomide in Multiple Myeloma Patients in Complete or Near Complete Remission
Brief Title: Allogeneic Myeloma GM-CSF Vaccine With Lenalidomide in Multiple Myeloma Patients in Complete or Near Complete Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Celgene (Industry); Aduro Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J16118; IRB00112179 (Other: JHM IRB)
Record Dates: First submitted 2017-11-30; First posted 2017-12-18 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; M-spike negative; GVax; GM-CSF secreting myeloma vaccine; MRD positive
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: All patients will continue on a standard dose of lenalidomide. Patients on the myeloma vaccine arm will receive injections in addition to lenalidomide unless otherwise clinically indicated, or until progression. Patients on myeloma plus Prevnar vaccine arm will receive injections of both allogenic myeloma vaccine and Prevnar vaccine in addition to lenalidomide unless otherwise clinically indicated, or until progression. Patients on the myeloma vaccine placebo arm will receive myeloma vaccine placebo on the same schedule as allogeneic myeloma vaccine. If assigned to either of the two arms that do not include Prevnar, then patients will receive placebo in lieu of Prevnar on the same schedule. The placebo will be saline. All patients will be followed for a minimum of 3 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lenalidomide plus GM-CSF Vaccine plus Prevnar13 (Experimental): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Prevnar vaccine will be administered with the GM-CSF vaccine administration.
  Interventions: Biological: GM-CSF vaccine; Drug: Lenalidomide; Drug: Prevnar13
- Lenalidomide Only (Placebo Comparator): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment. Patients will also get placebo GM-CSF vaccine and placebo prevnar13. Placebo will be saline.
  Interventions: Drug: Lenalidomide; Other: Placebo Prevnar13; Other: Placebo GM-CSF Vaccine
- Lenalidomide plus GM-CSF Vaccine (Placebo Comparator): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Patients will also be administered a placebo prevnar13 vaccination. Placebo will be saline.
  Interventions: Biological: GM-CSF vaccine; Drug: Lenalidomide; Other: Placebo Prevnar13

INTERVENTIONS:
Biological: GM-CSF vaccine — Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Other Names: GVAX
  Arms: Lenalidomide plus GM-CSF Vaccine; Lenalidomide plus GM-CSF Vaccine plus Prevnar13
Drug: Lenalidomide — Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Other Names: Revlimid
Drug: Prevnar13 — Prevnar will be administered at the same time points as the GM-CSF vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine.
  Other Names: pneumococcal vaccine
  Arms: Lenalidomide plus GM-CSF Vaccine plus Prevnar13
Other: Placebo Prevnar13 — Saline will be used for placebo. Placebo prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
  Arms: Lenalidomide Only; Lenalidomide plus GM-CSF Vaccine
Other: Placebo GM-CSF Vaccine — Saline will be used for placebo. Each placebo vaccine will consist of three total intra-dermal injections on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Placebo injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each injection is approximately 0.7-0.8ml.
  Arms: Lenalidomide Only

SUMMARY:
This study seeks to determine whether addition of an allogeneic myeloma vaccine can augment clinical responses to lenalidomide in patients with near complete remission (nCR), or complete remission (CR) leading to a significant improvement in progression-free survival.This main objective of this study is to compare the 2-year progression free survival of patients with multiple myeloma in CR or nCR, treated with lenalidomide plus an allogeneic myeloma vaccine in combination with lenalidomide (with or without Prevnar vaccine) or versus placebo in combination with lenalidomide (control arm).

DETAILED DESCRIPTION:
This is a single institution, three- arm, randomized controlled, Phase II study examining the clinical efficacy of an allogeneic GM-CSF secreting myeloma vaccine in combination with lenalidomide (with or without Prevnar) compared to lenalidomide and placebo (control arm).

Patients enrolled in the study must have two disease measurements (including the last one) consistent with a near complete remission (M-spike negative with persistence of immunofixation), or complete remission (M-spike negative, negative immunofixation, and <5% clonal plasma cells on bone marrow) per criteria for response in a 3 month period. All patients must be minimal residual disease (MRD) positive by NGS sequencing at enrollment.

Prior to enrollment, patients will have been treated with a lenalidomide containing regimen for a minimum of 6 cycles. All patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.

Patients will be randomized to receive either an allogeneic myeloma vaccine and Prevnar vaccine in combination with lenalidomide, or allogeneic myeloma vaccine without Prevnar vaccine in combination with lenalidomide, or lenalidomide in combination with placebo. Patients will receive allogeneic myeloma vaccine or placebo injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter for up to 3 years. If assigned to allogeneic myeloma vaccine plus Prevnar vaccine arm, Prevnar-13 will be administered with each allogeneic myeloma vaccine. If assigned to either of the two arms that do not include Prevnar, then patients will receive a placebo in lieu of Prevnar on the same schedule. All patients will be followed for a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma eligibility criteria are the following:
* Near complete remission (nCR) for ≥ 3 months defined as no measurable M-spike, and a positive serum immunofixation

  * For patients with a light chain only myeloma, they will be in deemed to be in a CR if they meet criteria for CR by International Myeloma Working Group (IMWG) consensus criteria 2016.
  * For patients with a light chain only myeloma that meet criteria for Very Good Partial Response (VGPR) by IMWG consensus criteria 2016 and are IFE -ve (negative serum immunofixation), they will be considered to be in a near complete remission (nCR).
* Or complete remission (CR) (no measurable M-spike, immunofixation negative and bone marrow plasma cells <5%)
* NDMM or RMM in nCR or CR having completed a minimum of 6 cycles of a lenalidomide based regimen for a minimum of ≥ 3 months
* NDMM or RMM a patients who have been off corticosteroids for ≥ 4 weeks
* Patients with NDMM or RMM who have had autologous stem cell transplant are eligible, but must be ≥ 12 months from transplant
* All patients must be MRD positive at 10-4 or greater by NGS sequencing at enrollment
* All patients must be currently taking Revlimid at screening.
* Age >18 years
* ECOG performance scores 0-2
* History of measurable serum or urine M protein or free light chains
* Life expectancy greater than 12 months
* Corrected serum calcium < 11 mg/dL, and no evidence of symptomatic hypercalcemia
* Serum creatinine< 2 mg/dl
* ANC >1000/µL
* Platelet >100,000/µL
* Total bilirubin <= 1.5 x ULN
* AST (SGOT) and ALT (SGPT) <= 3 x ULN.
* Ability to comprehend and have signed the informed consent.
* Have previously agreed to continue on maintenance therapy with lenalidomide concurrent with vaccine administration until disease progression, or clinical indication to cease therapy.
* Disease free of prior malignancies for at least 5 years with exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the uterus, cervix or breast.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to starting lenalidomide with each cycle (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Able to take prophylactic anticoagulation (aspirin 81 or 325 mg/daily or, for patients intolerant to ASA, warfarin or low molecular weight heparin).

Exclusion Criteria:

* Disease progression after stopping corticosteroids as defined as the appearance of a detectable serum or urine M-spike, or an absolute increase of >10 mg/dl between involved and uninvolved light chains, in the absence of measurable serum or urine M-protein .
* Patients who are MRD negative by NGS at screening.
* Patients with a known diagnosis of POEMS syndrome, plasma cell leukemia, CNS involvement, non-secretory myeloma and amyloidosis
* High-risk myeloma defined by presence of at least one of the following defining features on initial diagnostic, or most recent bone marrow biopsy:
* High risk chromosomal translocations by FISH: t(4;14), t(14;16), t(14;20),
* del(17p), del(1p), amplification 1q.;
* MyPRS GEP-70 high risk signature either from diagnosis or at time of registration for the study;
* LDH > 300 U/L at diagnosis;
* Relapse from prior therapy within 12 months.
* HIV disease, active infection requiring treatment with antibiotics, anti-fungal or anti-viral agents within 2 weeks of enrollment would be excluded from the study.
* Patients who have participated in any clinical trial, within the last four weeks, which involved an investigational drug.
* History of an active malignancy other than myeloma
* Autoimmune disease requiring active treatment.
* Known contra-indication to any component of allogeneic myeloma vaccine
* History of an allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed A Ali, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 participants were consented. 16 were screen failures. 8 participants were assigned to the arms.
Groups:
- Lenalidomide Plus GM-CSF Vaccine (Arm A): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Patients will also be administered a placebo prevnar13 vaccination. Placebo will be saline.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Placebo Prevnar13: Saline will be used for placebo. Placebo prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
- Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Prevnar vaccine will be administered with the GM-CSF vaccine administration.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Prevnar13: Prevnar will be administered at the same time points as the GM-CSF vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine.
- Lenalidomide Only (Arm C): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment. Patients will also get placebo GM-CSF vaccine and placebo prevnar13. Placebo will be saline.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Placebo Prevnar13: Saline will be used for placebo. Placebo prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
  Placebo GM-CSF Vaccine: Saline will be used for placebo. Each placebo vaccine will consist of three total intra-dermal injections on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Placebo injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each injection is approximately 0.7-0.8ml.
Period: Overall Study
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Started | 3 | 4 | 1
Completed | 3 | 3 | 1
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected for 8 participants
Groups:
- ARM A - Lenalidomide + GM-CSF Vaccine + Placebo Prevnar13: Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Patients will also be administered a placebo prevnar13 vaccination. Placebo will be saline.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Placebo Prevnar13: Saline will be used for placebo. Placebo Prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
- ARM B - Lenalidomide + GM-CSF Vaccine + Prevnar13: Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Prevnar vaccine will be administered with the GM-CSF vaccine administration.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Prevnar13: Prevnar will be administered at the same time points as the GM-CSF vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine.
- ARM C - Lenalidomide Only + Placebo GM-CSF Vaccine + Placebo Prevnar13: Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment. Patients will also get placebo GM-CSF vaccine and placebo prevnar13. Placebo will be saline.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Placebo Prevnar13: Saline will be used for placebo. Placebo prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
  Placebo GM-CSF Vaccine: Saline will be used for placebo. Each placebo vaccine will consist of three total intra-dermal injections on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Placebo injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each injection is approximately 0.7-0.8ml.
- Total: Total of all reporting groups
Arm/Group | ARM A - Lenalidomide + GM-CSF Vaccine + Placebo Prevnar13 | ARM B - Lenalidomide + GM-CSF Vaccine + Prevnar13 | ARM C - Lenalidomide Only + Placebo GM-CSF Vaccine + Placebo Prevnar13 | Total
Number analyzed (Participants) | 3 | 4 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 0 | 3
  >=65 years | 2 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 2 | 3 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 3 | 2 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression Free Survival
Description: Number of participants without disease progression at 2 years.
Time Frame: 2 years
Population: Evaluable patients at 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm A): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Prevnar vaccine will be administered with the GM-CSF vaccine administration.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Prevnar13: Prevnar will be administered at the same time points as the GM-CSF vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine.
- Lenalidomide Plus GM-CSF Vaccine (Arm B): Patients will continue on a standard dose of lenalidomide as a single agent until progression, or treatment limiting toxicity, following enrollment.
  Patients assigned to vaccine therapy will receive injections on day 14 (+/-3 days) of cycles 1, 2, 3 and 6 from enrollment, and then annually thereafter. Patients will also be administered a placebo prevnar13 vaccination. Placebo will be saline.
  GM-CSF vaccine: Each vaccination will consist of three total intra-dermal injections, on day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). In the event that the specified limb is contraindicated, the dominant arm may be used. Vaccine injection sites shall be at least 5 cm at needle entry from the nearest neighbor. The approximate volume of each vaccination injection is approximately 0.7-0.8ml.
  Lenalidomide: Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5-25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Placebo Prevnar13: Saline will be used for placebo. Placebo prevnar will be administered at the same time points as the GM-CSF vaccine or Placebo GM-CSF Vaccine (day 14 of cycles 1, 2, 3, 6 and annually for a minimum of 36 months), but on the opposite arm from GM-CSF vaccine or placebo GM-CSF vaccine.
Arm/Group | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm A) | Lenalidomide Plus GM-CSF Vaccine (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 3 | 3 | 1
Participants | 3 | 3 | 1

2. Secondary Outcome: Response Conversion Rate
Description: Number of participants who converted from near complete remission (nCR) to complete remission (CR) as measured by the International Myeloma Working Group Uniform Response Criteria. Near complete remission is defined as negative serum and urine electrophoresis, < 5% plasma cells in the bone marrow, and positive serum and/or urine immunofixation. Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
Time Frame: 2 years
Population: Patients evaluable at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 0

3. Secondary Outcome: MRD Conversion Rate
Description: Number of participants who convert from MRD (Minimal Residual Disease) positive status to MRD negative status as determined through next generation sequencing (NGS).
Time Frame: 2 years
Population: Patients who were evaluable at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 0

4. Secondary Outcome: Time to Response
Description: Median time for conversion of response from near complete remission (nCR) to complete remission (CR) as measured by the International Myeloma Working Group Uniform Response Criteria. Near complete remission is defined as negative serum and urine electrophoresis, < 5% plasma cells in the bone marrow, and positive serum and/or urine immunofixation. Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells as measured by immunofixation converting from positive to negative.
Time Frame: 2 Years
Population: No participants reached response conversion from near complete remission to complete remission.
Measure: Median (Full Range); unit: days
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 3 | 3 | 1
days | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of months without disease progression.
Time Frame: 3 and 5 years
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Evaluate Toxicity of Allogenic Myeloma Vaccine
Description: Number of participants experiencing adverse events grade 3 or higher, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Time Frame: 3 years
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Measure Tumor Specific Immunity and Correlate With Systemic Immunity
Time Frame: 3 years
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Lenalidomide Plus GM-CSF Vaccine (Arm A) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm B) | Lenalidomide Only (Arm C)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment up to 2 years
Arm/Group | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm A) | Lenalidomide Only (Arm C) | Lenalidomide Plus GM-CSF Vaccine (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide Plus GM-CSF Vaccine Plus Prevnar13 (Arm A) (N=3) | Lenalidomide Only (Arm C) (N=4) | Lenalidomide Plus GM-CSF Vaccine (Arm B) (N=1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Basal cell, nose (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was significantly negatively impacted by COVID pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03376477/Prot_SAP_000.pdf